CLINICAL TRIAL: NCT06601088
Title: Acute Achilles Tendon Rupture - Intervention With Neuromuscular Electrical Stimulation
Brief Title: Achilles Tendon Rupture - Intervention With Electrical Stimulation
Acronym: C-NMES-ATR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Paul Ackermann, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C-NMES-ATR
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Achilles Tendon Ruptures; Immobilization; Venous Thromboembolism (VTE); Muscle Atrophy
Keywords: neuromuscular electrical stimulation; duplex ultrasound
MeSH Terms: conditions — Venous Thromboembolism; Muscular Atrophy | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group with standard lower-limb immobilization (No Intervention): The control group will be treated according to the standard regimen with a lower limb immobilization in a stable orthosis during eight weeks.
- Intervention group with additional Neuromuscular Electrical Stimulation' (Experimental): The intervention group will during the eight weeks lower limb immobilization receive an additional intervention with calf Neuromuscular Electrical Stimulation (C-NMES) underneath the orthosis.
  Interventions: Device: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — Patients will be instructed to apply the wearable NMES-therapy continuously, both day and night at least 10h/daily.
  Other Names: Electrical Stimulation; NMES; C-NMES
  Arms: Intervention group with additional Neuromuscular Electrical Stimulation'

SUMMARY:
Acute Achilles tendon rupture (ATR) is an injury that is commonly associated with complications, such as blood clotting, muscle loss and tendon lengthening, all of which affect the long-term outcome and return to sports. These complication are related to the treatment of ATR with lower leg immobilization in a boot.

The investigators aim to demonstrate that an intervention with calf neuromuscular electrical stimulation (C-NMES) during leg immobilization after ATR can 1) reduce blood clots, 2) lower the degree of muscle loss, 3) decrease tendon lengthening and 4) improve long-term outcome.

DETAILED DESCRIPTION:
The participants will be divided by chance into two separate groups that compare standard treatment (control group) with C-NMES in addition to standard treatment (intervention group).

A total of 220 patients with diagnosed ATR will be included. The control group will be treated according to the standard regimen with a lower leg immobilization in a stable orthosis during eight weeks. The intervention group will during the eight weeks lower limb immobilization receive an additional intervention with C-NMES underneath the orthosis.

The total number of blood clots, venous thromboembolism incidence, up to mobilization, is defined as deep venous thrombosis (leg blood clots) assessed by screening duplex ultrasound, or pulmonary embolism (lung blood clots). Calf muscle loss, tendon length, and weight-bearing, will be studied at two and eight weeks. At six weeks and 12 months, validated self-reported function (ATRS) and self-reported health, return to sports, calf muscle function, and tendon length will be recorded for comparison between the two treatment groups. Secondary outcomes are coagulation factors, healing biomarkers and cardiovascular biomarkers.

The results of this study should contribute to an improved treatment regimen after ATR that allows for a safer and quicker return to activity and sports. Adjuvant NMES can readily be implemented in daily healthcare to lower complication risks, improve healing, reduce healthcare costs and improve return to sports.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute unilateral Achilles tendon rupture
* Included within 10 days after injury.

Exclusion Criteria:

* Inability to give consent to participate,
* ongoing treatment with anticoagulants,
* known allergy to contrast agents,
* planned follow-up at another hospital,
* inability to follow instructions,
* known renal failure,
* heart failure with pitting edema,
* thrombophlebitis,
* thromboembolic disease within the last 3 months,
* previous surgery of the tendon,
* known malignancy,
* hemophilia,
* pregnancy,
* treatment with high doses of acetylsalicylic acid.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Venous thromboembolic events (VTE) | 8 weeks
  VTE, is defined as symptomatic/ asymptomatic DVT assessed at the end of immobilization, i.e. 8 weeks, by compression duplex ultrasound (CDU) screening, or symptomatic pulmonary embolism detected by computer tomography. Assessors of CDU will be skilled ultrasonographists, masked to the treatment allocation. The CDU-examination will document absence/presence of thrombus in the calf, popliteal and femoral veins separately

SECONDARY OUTCOMES:
Patient function | 12 months
  Functional evaluation of healing will be performed by the validated heel-rise test at one-year post-injury.
Callus production | 8 weeks
  Callus production will be assessed at eight weeks using microdialysis followed by quantification of procollagens for tendon healing.
Treatment adherence | 8 weeks
  Treatment adherence to allocated treatment, NMES, will be registered by the patient and by the device.
Adverse events | 8 weeks
  Adverse events that will be registered are 1) Any damage to the skin of the legs including infection. 2) Any reasons for prematurely stopping the NMES. 3) Any fall associated with significant injury occurring within 6 weeks of enrollment. The frequency of the adverse events of each group will be presented.
Fasting blood glucose | 8 weeks
  Fasting blood glucose will be assessed at inclusion and at eight weeks. A fasting blood sugar level less than 100 mg/dL (5.6 mmol/L) will be considered normal. A fasting blood sugar level from 100 to 125 mg/dL (5.6 to 6.9 mmol/L) will be considered considered prediabetes. If it is 126 mg/dL (7 mmol/L) or higher it will be considered diabetic.
Cholesterol levels | 8 weeks
  Will be assessed at inclusion and at eight weeks. Total cholesterol less than 200 Mmol/l will be considered good. Total cholesterol 200-239 Mmol/l will be considered moderately elevated. Total cholesterol 240 Mmol/l or higher will be considered high.
Blood pressure | 8 weeks
  Systolic blood pressure less than 120 mmHg and diastolic blood pressure less than 80 mmHg will be considered optimal.
  Systolic blood pressure between 120-129 mmHg and diastolic blood pressure between 80-84 mmHg will be considered normal.
  Systolic blood pressure between 130-139 mmHg and diastolic blood pressure between 85-89 mmHg will be considered slightly high.
  Systolic blood pressure greater or equal to 140 mmHg and diastolic blood pressure greater or equal to 90 mmHg will be considered high.
Muscle atrophy | 12 months
  At 2 and 6 weeks and 6 and 12 months postoperatively, B-mode ultrasound imaging will be performed to assess the cross-sectional area (CSA) of the Achilles tendon, the gastrocnemius CSA, as well as the thickness of soleus. The injured and healthy sides will be compared.
Tendon lengthening | 12 months
  At 2 and 6 weeks and 6 and 12 months postoperatively, B-mode ultrasound imaging will be performed to assess the length of the Achilles tendon. The injured and healthy sides will be compared. A larger difference between the sides will be considered a worse outcome.
Patient-reported outcome - ATRS | 12 months
  The validated Achilles Tendon total Rupture Score (ATRS) will be assessed at 6 and 12 months. [0-100, a higher score mean a better outcome].
Patient-reported outcome - EuroQol (EQ-5D-5L) | 12 months
  The validated EuroQol (EQ-5D-5L), will be assessed at 6 and 12 months. [A five-digit code will be generated, where each digit will be between 1-5, a lower digit in each position mean a better outcome in that dimension]. The five-digit code will generate an index between 0-1, where a lower value is worse outcome. The index will be compared with a country specific index.
Blood-flow quantification | 8 weeks
  VTE-preventive mechanisms will be analyzed at the eight week visit by assessments by blood-flow quantification using ultrasound. Peak popliteal/femoral blood velocity (cm/second) will be calculated using custom ultrasound software.
Coagulation factors | 8 weeks
  VTE-preventive mechanisms will be analyzed at the baseline and eight week visit by assessments of coagulation factors. Overall hemostatic potential (OHP), D-dimer, endogen trombin potential, fibrinogen, trombin antitrombin complex, plasmin antiplasmin complex, will be assessed in blood samples. The percentage increase/decrease between baseline and eight weeks assessment will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ackermann, Prof,MD,PhD, Principal Investigator — Karolinska Institutet and Karolinska University Hospital

IPD SHARING:
Plan to Share IPD: Yes
On reasonabe request data will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: June 2025 and will be available 2 years
Access Criteria: On reasonabe request data will be shared.

REFERENCES:
- [Background] Alharbi A, Li J, Womack E, Farrow M, Yarar-Fisher C. The Effect of Lower Limb Combined Neuromuscular Electrical Stimulation on Skeletal Muscle Signaling for Glucose Utilization, Myofiber Distribution, and Metabolic Function after Spinal Cord Injury. Int J Environ Res Public Health. 2023 Oct 21;20(20):6958. doi: 10.3390/ijerph20206958. PMID 37887696
- [Background] Hajibandeh S, Hajibandeh S, Antoniou GA, Scurr JR, Torella F. Neuromuscular electrical stimulation for the prevention of venous thromboembolism. Cochrane Database Syst Rev. 2017 Nov 21;11(11):CD011764. doi: 10.1002/14651858.CD011764.pub2. PMID 29161465
- [Background] Aufwerber S, Heijne A, Edman G, Silbernagel KG, Ackermann PW. Does Early Functional Mobilization Affect Long-Term Outcomes After an Achilles Tendon Rupture? A Randomized Clinical Trial. Orthop J Sports Med. 2020 Mar 16;8(3):2325967120906522. doi: 10.1177/2325967120906522. eCollection 2020 Mar. PMID 32206673
- [Background] Aufwerber S, Svedman S, Silbernagel KG, Ackermann PW. Long-term patient outcome is affected by deep venous thrombosis after Achilles tendon rupture repair. Knee Surg Sports Traumatol Arthrosc. 2024 Aug;32(8):2184-2193. doi: 10.1002/ksa.12240. Epub 2024 May 26. PMID 38796725
- [Background] Svedman S, Marcano A, Ackermann PW, Fellander-Tsai L, Berg HE. Acute Achilles tendon ruptures between 2002-2021: sustained increased incidence, surgical decline and prolonged delay to surgery-a nationwide study of 53 688 ruptures in Sweden. BMJ Open Sport Exerc Med. 2024 Jul 18;10(3):e001960. doi: 10.1136/bmjsem-2024-001960. eCollection 2024. PMID 39040046